CLINICAL TRIAL: NCT00106457
Title: 20 Year Changes in Fitness & Cardiovascular Disease Risk - Ancillary to CARDIA
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1290; R01HL078972-04 (NIH)
Record Dates: First submitted 2005-03-24; First posted 2005-03-25 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-11

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Metabolic Syndrome X; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Metabolic Syndrome; Hypertension; Obesity

SUMMARY:
To understand the complex, longitudinal relations between physical fitness, physical activity, body mass and composition and fat distribution, and genetic factors and their independent or interactive effects on the development of obesity, the metabolic syndrome, and sub-clinical cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Although an age-related decline in aerobic capacity is well documented, the impact of physical activity, body fat, and genetic variation on the rate of change is not well understood. In addition, little is known about how rate of change in aerobic capacity during early and middle adulthood affects the development of cardiovascular disease risk factors or the incidence of subclinical and clinical cardiovascular disease (CVD) related end-points. The study addresses these issues by conducting an ancillary study in conjunction with the Year 20 CARDIA (Coronary Artery Risk Development in Young Adults) examination, which is scheduled to take place beginning in June, 2005. Approximately 3,650 (75%) of the surviving members of the initial cohort of African American and white men and women will return for the Year 20 exam, at which point they will be 38-50 years old.

CARDIA is a National Heart, Lung, and Blood Institute-supported longitudinal study which measures changes in coronary heart disease risk factors in cohorts of Black and white males and females who were 18 to 30 years of age at baseline. Also, the study identifies life styles during this age span which influence these changes in risk factors.

DESIGN NARRATIVE:

The overall goal of the ancillary study is to understand the complex, longitudinal relations between physical fitness, physical activity, body mass and composition and fat distribution, and genetic factors and their independent or interactive effects on the development of obesity, the metabolic syndrome, and sub-clinical CVD. To accomplish this goal, all Year 20 CARDIA participants will be measured for: 1. Aerobic capacity, by means of a symptom-limited graded exercise treadmill test, using the same protocol as that used in CARDIA at the Year 0 and Year 7 exams; 2. Body composition and fat distribution, using a whole body dual energy x-ray absorptiometery (DEXA) scan; 3. Physical activity, using 7 days of accelerometer recordings; and 4. DNA sequence variants in selected candidate genes associated with cardiorespiratory fitness, components of the metabolic syndrome, and response to regular exercise, using stored DNA.

Data from this ancillary study will be combined with core CARDIA examination data to address the following aims: a. Examination of the contribution of body mass and composition, fat distribution, objectively measured physical activity and specific genetic polymorphisms to the variance in Year 20 aerobic capacity and in age-related decline in aerobic capacity over a 20-year time period from young adulthood to mid-life, stratifying by race and gender. b. Longitudinal examination of the effect of aerobic capacity on changes in cardiovascular disease risk factors and on the incidence of CVD-related endpoints (e.g. hypertension, metabolic syndrome, subclinical disease [e.g. coronary artery calcium]).

ELIGIBILITY:
No eligibility criteria

Ages: 38 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sidney — Kaiser Foundation Research Institute

REFERENCES:
- [Derived] Shikany JM, Jacobs DR Jr, Lewis CE, Steffen LM, Sternfeld B, Carnethon MR, Richman JS. Associations between food groups, dietary patterns, and cardiorespiratory fitness in the Coronary Artery Risk Development in Young Adults study. Am J Clin Nutr. 2013 Dec;98(6):1402-9. doi: 10.3945/ajcn.113.058826. Epub 2013 Oct 2. PMID 24088719